CLINICAL TRIAL: NCT04837222
Title: Observational, Non-interventional, Multicenter Study Aimed at Collecting Prospective Data Related to Study Safety and Effectiveness in Real Clinical Practice in Patients With CD30+ Lymphoma (BRAVE Study)
Brief Title: A Study of Brentuximab Vedotin in Adults With CD30-positive Lymphoma
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C25022; U1111-1258-8445 (Registry Identifier: WHO)
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with CD30-positive Lymphoma: All participants diagnosed with CD30-positive lymphoma who are receiving or will recieve brentuximab vedotin will be observed prospectively over 24-month period, unless withdrawal of informed consent, lost or death, whichever comes first.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
Participants with CD30-positive lympoma will be treated with brentuximab vedotin according to their clinic's standard practice.

The main aim of this study is to collect information on any side effects from treatment with brentuximab vedotin. Other aims are to collect information on how brentuximab vedotin is used to treat these participants and the outcomes of these participants.

DETAILED DESCRIPTION:
This is an observational, non-interventional, prospective study in participants with CD30-positive lymphoma who are receiving or will receive the standard treatment of brentuximab vedotin. This study will assess the safety profile and effectiveness of brentuximab vedotin in the real-world clinical practice.

The study will enroll approximately 1000 participants. The data will be collected and recorded in the medical record for the purpose of medical care and also recorded in electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

• All participants with CD30-positive lymphoma

This multi-center trial will be conducted in China. All participants will be followed up for 24 months unless withdrawal of Informed Consent, lost or death, whichever comes first. The overall duration of the study will be approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing treatment with brentuximab vedotin (of less than 3 months from initial treatment with brentuximab vedotin) or to be received with brentuximab vedotin.
2. CD30-positive lymphoma by INV (any CD30 expression)

Exclusion Criteria:

1. Who currently participates in or with plan to participate in any interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CD30-positive lymphoma, who have been prescribed brentuximab vedotin in clinical practice will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting one or More Serious Adverse Events (SAEs) | Up to 4 years

SECONDARY OUTCOMES:
Number of Participants Reporting one or More Adverse Events (AEs) | Up to 4 years
Number of Participants Reporting one or More Adverse Drug Reactions (ADRs) | Up to 4 years
  ADRs refers to AE related to administered drug.
Number of Participants With Dose Adjustments During the Study | Up to 4 years
Number of Participants Based on Usage of Brentuximab Vedotin | Up to 4 years
Number of Cycles of Brentuximub Vedotin Administered in Routine Clinical Practice | Up to 4 years
Number of Participants Based on Disease Characteristics | Up to 4 years
  Number of participants will be reported based on the type of lymphoma, stage, lines of therapy.
Time to Next Treatment (TTNT) | From start of each line of therapy until next line of therapy (up to 4 years)
  TTNT is defined as time between start of each line of a therapy to the next line of therapy.
Objective Response Rate (ORR) | Up to 4 years
  ORR is defined as the percentage of participants with complete response (CR) and partial response (PR) after treatment in the total number of assessable cases.
Duration of Response (DOR) | From date of first documented CR until PD (up to 4 years)
  DOR is calculated from the time of documentation of a CR to documentation of disease progression. CR is defined as disappearance of all residual disease and tumor lesions. Disease progression (PD) is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Progression Free Survival (PFS) Rate | 1 year and 2 years
  PFS rate is calculated as the percentage of participants who reported PFS (at 1st year, 2nd year) as per investigator's assessment after brentuximab vedotin treatment.
Overall Survival (OS) Rate | 1 year and 2 years
  OS rate is measured as the percentage of participants who reported death (at 1st year, 2nd year) after brentuximab vedotin treatment.
Change From Baseline in Quality of Life (QoL) Assessed Using Functional Assessment of Cancer Therapy Lymphoma (FACT-Lym) Questionnaire Version 4 | Up to 4 years
  The FACT-Lym questionnaire is a validated instrument for assessing the impact of lymphoma on health related quality of life and contains 42 questions covering health related quality of life, common lymphoma symptoms, and treatment side-effects. It contains four core subscales including: Physical Wellbeing, Social/Family Wellbeing, Emotional Wellbeing, and Functional Wellbeing. All questions are answered on a 5-point likert scale ranging from 0 to 4: 0=not at all,1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. Higher scores are associated with a better quality of life.
Cost-effectiveness Ratio | Up to 4 years
  Cost-effectiveness ratio will be assessed by the direct cost (including medication, injunction, test, nursing fee, etc.) under brentuximab vedotin treatment divided by the total percent of CR and PR.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- China (31):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospita, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - ZhuJiang Hosptital of Southern Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - HenanProvincial CancerHospital, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hodpital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - ShandongProvincial CancerHospital, Jinan, Shandong
  - Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - ShanxiProvincial CancerHospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Yunnan First People's Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/60749a78688ad8001f42fb91??page=1&idFilter=C25022